CLINICAL TRIAL: NCT06170112
Title: Evaluation Of The Effect Of Spinal Orthosis On Tactile Sense And Balance In Individuals With Lumbal Curve And Adolescent Idiopathic Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Başak İŞÇİOĞLU, Orthosist Prosthetist, Istanbul Medipol University Hospital
Other Study IDs: Orthosis Prosthesis
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; Sense of Touch; Dynamic balance; Spinal orthosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Orthosis: There are pressure forces applied by the design of the spinal orthosis in changing the biomechanics of the scoliotic spine. In the design of the spinal orthosis designed with the 3-point principle, there is a corrective lateral force applied to the main curvature area and two support forces opposing this force. There are breathing spaces in the back area.
  Interventions: Other: Spinal Orthosis Application

INTERVENTIONS:
Other: Spinal Orthosis Application — Spinal orthosis treatment is to prevent secondary curvature and provide correction. Corrective pressure forces in spinal orthosis are basically; There are pressure points on the material of the spinal orthosis, pressure pads, and velcros used to adjust the tightness and ensure the stability of the orthosis. The duration of use of spinal orthoses varies from patient to patient; It is known that using it for an average of 23 hours a day gives the best results. Orthosis use is required for 12 weeks during the study.

SUMMARY:
In individuals with lumbar curvature, significant regressions in the curvature have been observed with spinal orthosis treatment, especially with use of a minimum of 20 hours a day. Symptoms such as numbness and decreased sense of touch are observed in the areas where the curvature is located, and changes in the skin structure are affected by the changes in the spine. Sensory testing may vary with changes in body posture. At the same time, the use of spinal orthosis, balance, fat mass, and the presence of pain show us sensitivity to touch on the skin. Sensory stimuli on the skin and trunk posture are interconnected. There are a limited number of studies in the literature examining the effects of sensory test results and fat mass on individuals diagnosed with AIS after using a spinal orthosis.

DETAILED DESCRIPTION:
The purpose of this study is to examine how spinal orthoses affect lumbar curvature, tactile sensation, dynamic balance, skinfold thickness, and quality of life in people with adolescent idiopathic scoliosis. The 40 participants in the study will be between the ages of 10 and 18, with Cobb angles ranging from 20 to 45 degrees.Consent forms will be obtained from all participants and parents participating in the study.

Semmes Weinstein Monofilament kit will be used to measure participants' sense of touch, Skinfold Caliper to measure subcutaneous fat tissue, Y-Balance Test for Dynamic Balance, and Scoliosis Research Society 22 (SRS-22) Evaluation Questionnaire. Measurements will be recorded before the birth of the corset and 12 weeks after the start of corset use. At the end of the 12th week, the brace will be evaluated for satisfaction with the Brace Questionnaire (BRQ).

Socio- demographic form information will be given at the first interview. In addition to the anamnesis, this form includes questions about whether the person exercises or not, whether there is a family member diagnosed with scoliosis, and the doctor's instructions for use of the orthosis.

Sense of Touch Assessment- Semmes Weinstein Monofilament Kit will be used in the study. This test is one of the tests commonly used to evaluate light touch sensation. Although it is mostly used in the palmar area, it is also used in certain parts of the body to test light touch sensation. Semmes-Weinstein Monofilament test is performed using filaments of different diameters with the same length. The thicknesses of the filaments are 2.83, 3.22, 3.61, 3.84 and 4.31. As the filament diameter thickens, the pressure given and the sensory input given increase accordingly. In the study, in individuals diagnosed with adolescent idiopathic scoliosis and with lumbar curvature, these filaments will be applied to two different regions of the curvature, concave and convex, at T10, L4 and L5, in order from thinnest to thickest. The number of the first monofilament felt will be recorded. Pressure will be applied until the 2.83 mm monofilament, which has the thinnest diameter, is curled, the person will be asked whether he/she feels the pressure, and if not, the application will continue by increasing the filament thickness accordingly.

Fat Tissue Measurement- Skinfold Caliper thickness measurement is performed to determine the fat tissue under the skin. A significant part of the fat in the body is collected under the skin. The thickness of the skinfold is evaluated with a special caliper called skinfold. Measurement is made by holding the skin and subcutaneous tissue with the thumb and index finger and pulling the natural skin piece away from the muscle. It is read in millimeters from the caliper indicator. Measurement of the evaluated area should be done twice, and if the difference is more than 2 mm, the measurement should be repeated. The body parts measured can be listed as triceps, biceps, subscapula, suprailiaca, front of the thigh, inner side of the calf, abdomen, chest and midaxilla. It is known that low body fat is a risk factor for the onset of scoliosis. In our study, fat tissue measurements will be made in the axilla, abdominal, suscapular and suprailiac regions.

Dynamic Balance- Y Balance Test After the foot of the party to be tested is placed behind the red line on the platform, they will be asked to push the distance indicator in all three directions (anterior, postromedial and posterolateral) as far as possible with the foot in the air. After two trials are made in each direction before the test, three measurements will be taken for each direction during the test phase. For each direction, the total score obtained by dividing the best value of the three maximum distances by the leg length and multiplying by 100 will be calculated and noted. The test will be terminated when the person lifts the heel of the tested foot standing on the platform to maintain balance during the test, loses contact with the distance indicator, uses it as support to restore the lost balance and cannot return to the starting position.

Scoliosis Research Society's Health-related Quality of Life- 22 (SRS-22) survey form; It is a quality of life questionnaire created specifically for individuals diagnosed with scoliosis. It includes parameters of pain, self-appearance, function-activity, mental health, and satisfaction with treatment. It also has a role in evaluating changes within treatment. It will be filled in by the researcher together with the patient. It will be calculated by giving an answer value to all 22 questions within a 5-point indicator chart. Each statement has responses ranging from negative to positive. The most negative answer will be scored as 1 point and the most positive answer will be scored as 5 points. All questions will be evaluated under the total result score.

Brace Questionnaire (BRQ)- Recording the evaluation of brace treatment and the feedback from the patient gives the clinician objective information about choosing the right treatment method. It consists of 34 questions grouped under 8 main headings. The domains include general health perception, physical functioning, emotional functioning, self-confidence and aesthetics, vitality, school activity, body pain, and social functioning. The score of each question (between 1 and 5) is multiplied by 20 to reach the final score, and higher scores indicate a better quality of life. Since it questions the effect of corset use on many parameters in a versatile way, it offers us an idea about the quality of life with corset in a practical and easy way.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Adolescent Idiopathic Scoliosis (AIS) between the ages of 10-18,
* Curvature only in the lumbar region,
* 20-45 degree curvature degree,
* Being deemed suitable for spinal orthosis use by the doctor,
* Not having used a spinal orthosis before

Exclusion Criteria:

* Having different diagnoses such as congenital scoliosis, spina bfida, traumatic scoliosis, osteoporosis,
* Having had spine surgery
* Having used a scoliosis spinal orthosis,
* Having an accompanying disease that may prevent the use of spinal orthosis and
* Failure to sign the consent form required to participate in the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals between the ages of 10-18 who have been diagnosed with AIS by a doctor come to our clinic. Following clinical evaluations, a spinal orthosis evaluation will be performed. Individuals must not have used a spinal orthosis before.They should not have any accompanying neurological disease.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-03-06 (Estimated)

PRIMARY OUTCOMES:
The effect of spinal orthosis on the sense of touch | 5 minute
  Individuals between the ages of 10-18 included in the study will touch the ends of the monofilament kit, consisting of 6 different tips, to the concave and convex sections of the slope in the T10-L4 and L5 regions. The results are recorded when the individual answers "I felt it/I didn't feel it". Evaluations will be made immediately before orthosis use and 12 weeks after orthosis use.

SECONDARY OUTCOMES:
Effect of spinal orthosis on dynamic balance | 10 minute
  The lower extremity to be evaluated is lifted onto the testing platform. It is desired to extend to the anterior, posterolateral and posteromedial directions, respectively. The longest distance it can reach is recorded.
Effect of spinal orthosis on fat tissue | 5 minute
  The midaxilla, abdomen, subscapular and suprailiac regions to be evaluated are compressed with the thumb and index finger, and the collected skin piece is measured with a caliper.
The effect of spinal orthosis on quality of life | 20 minute
  A survey is conducted to monitor individuals' spinal orthosis and health-related quality of life during the period of spinal orthosis use.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Iscioglu, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No